CLINICAL TRIAL: NCT05895760
Title: Effectiveness of a Multi-component Physical Exercise Online on Physical Performance in Community-dwelling Older Adults: a Randomized Controlled Trial
Brief Title: Effectiveness of a Multi-component Physical Exercise Online
Acronym: MEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Iberoamericana A.C., Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SALUD-2021-PHYSICAL EXERCISE; 35/2020 (Registry Identifier: Ejercicio multicomponente para mejorar el desempeño físico)
Record Dates: First submitted 2023-05-05; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Older Adults
Keywords: older adults; multi-component physical exercise; online; physical performance

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial, including 110 older adults (68.45±5.54 years), were divided into two parallel groups: an MPE group (n = 55) and a control group (n = 55).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-component physical exercise online intervention (MPE) (Experimental): The exercise program included endurance, strength, coordination, balance, and flexibility exercises which were carried out for 3 months.
  Interventions: Other: Multi-component physical exercise online intervention
- Control group (No Intervention): The control group received educational sessions on health prevention related to physical exercise.

INTERVENTIONS:
Other: Multi-component physical exercise online intervention — A multicomponent exercise program was implemented consisting of a combined program of endurance, strength, coordination, balance, and flexibility exercises depending on the level of functional capacity.
  Three types of physical exercise programs were designed according to the physical performance level of each participant. The first type of exercise program training was performed for frail adults with an SPPB score of 4 to 6, the second was for the pre-frail adults with an SPPB score of 7 to 9 and the third for robust adults with an SPPB of 10 to 12.
  Arms: Multi-component physical exercise online intervention (MPE)

SUMMARY:
Objective: to assess the effectiveness of a multi-component physical exercise online intervention (MPE) on physical performance (PP) in community-dwelling older adults.

Methods: a randomized controlled trial, including 110 older adults (68.45±5.54 years), were divided into two parallel groups: an MPE group (n = 55) and a control group (n = 55). The exercise program included endurance, strength, coordination, balance, and flexibility exercises which were carried out for 3 months. The control group received educational sessions on health prevention related to physical exercise. The main endpoint was a change in PP assessed with the short physical performance battery (SPPB). It is also evaluated other variables such as sociodemographic (sex, age, education level), health conditions (cognitive impairment, polypharmacy, comorbidity, frailty, sarcopenia, depressive and anxiety symptoms), functional dependence through scales of activities of daily living (ADL), nutrition (risk of malnutrition, weight, height, body mass index (BMI), calf and waist circumference) and lifestyles (physical activity, alcoholism, and smoking). Comparisons were made in the follow-up measurements between groups by an independent t-test and baseline and follow-up measurements in both groups by a paired t-test.

DETAILED DESCRIPTION:
Methods Study design and participants. The study was a randomized controlled trial conducted from June to October 2021. The study population was randomly selected from the FraDySMex study (Frailty, Dynapenia and Sarcopenia in Mexican Adults), adults aged 50 years and older. The adults were residents of Mexico City from three different municipalities (Cuajimalpa, Álvaro Obregón and Magdalena Contreras). The protocol was approved by the Committee on Ethics in Research of the "Iberoamerican University, Mexico City. with No35/2020. Informed consent was obtained from each participant who signed it after fully understanding the procedures.

The eligibility criteria were the following:

* Adults 60 and over years
* Adults who had an electronic device with internet access for video calls.

The exclusion criteria were:

* Adults self-reported walking disability, with the inability to complete the short physical performance battery (SPPB)
* Adults with severe functional dependence (defined as a Barthel index ≤ 60/100 score)
* Adults with cognitive impairment (defined as a mini-mental state examination (MMSE) score <24/30)
* Adults with terminal illness
* Adults who were participation in a physical activity or nutritional program
* Adults with a limb loss or use of lower or upper limb prostheses
* Adults with a history of injuries (fractures/falls) of less than one year in hip, knee or ankle joints and with surgery in the last 6 months or contraindications to perform trial activities in the judgment of medical personnel.
* Adults who presented any medical condition or adverse symptoms during the intervention that made it impossible to carry out the physical exercise program
* Adults who did not keep three times consecutive were eliminated from the study.

Sample size estimate / power calculations The sample size calculation was based on the primary outcome SPPB with power of .80 [1-β], 2-sided α-error (95% CI), 2 groups, 2 measurements. One hundred participants were required in order to detect a clinically meaningful change of ≥1.0 point with a SD of 0.99 points. To account for potential dropouts before study completion, we will inflate the sample size by 10% losses during follow-up, resulting in a total sample size of 110 individuals (55 participants allocated to each group). With a sample of 1000 adults from the FraDySMex study, were selected 110 adults and they will be assigned to groups by computer random number generation and were assigned in 1:1 ratio (intervention group and control group). It was simple-blind, since the participants did not know which they were group. Figure 1 shows the population flow diagram.

Safety All study staff monitored participant safety and reported three categories of adverse events: serious adverse events, unexpected adverse events (those potentially related to study procedures or activities and not listed in the informed consent form or study protocol), and adverse events that occurred while the participant was under the supervision or guidance of study staff.

Interventions Intervention group. A multicomponent exercise program (MEP) was implemented consisting of a combined program of endurance, strength, coordination, balance, and flexibility exercises depending on the level of functional capacity (i.e. severe, moderate, and mild limitation). The recommendations of the ViviFrail project were followed to form the groups depending on their (short physical performance battery) SPPB score.

Three types of physical exercise programs were designed according to the physical performance level of each participant. The first type of exercise program training was performed for frail adults with an SPPB score of 4 to 6, the second was for the pre-frail adults with an SPPB (short physical performance battery) score of 7 to 9 and the third for robust adults with an SPPB of 10 to 12. The multi-component program was developed with the support of a physical training specialist, a medical rehabilitator, gerontological nutritionists and geriatrics. First, warm-up exercises, general exercises, and return-to-calm exercises were structured for each group an then videos were made to upload the exercise program on a YouTube plataform.

To start the intervention, a message was sent a few days beforehand to remind about the appointment and the materials for the corresponding session. The intervention for each of the participants was carried out individually through the Zoom app or by WhatsApp video call 3 times a week with the supervision of health professionals with a duration per session of 45-60 min. At the end of the session, the OMNI- RES physical exercise effort scale was applied, which has a score from 0 to 10, classified as 0 extremely easy to 10 extremely hard. In addition, the participant's physical fitness and physical activity status were monitored through a series of questions at the beginning of each week of intervention to ensure the older adult was able to continue with the intervention.

Control group This group was invited to remote meetings every 15 days in which education on exercise-related health prevention was provided. Topics such as: benefits of multicomponent exercise for older adults, recommendations for physical exercise training in older adults, recommendations for an active aging, healthy eating for older adults, my plate for older adults. The physical rehabilitator and gerontological nutritionists were in charge of providing the recommendations and the session lasted approximately. In addition, they were instructed not to participate in any physical exercise program during the study period and to continue with their usual activities.This information is available on the You Tube platform. https://www.youtube.com/@nutriciongeriatrica/videos

Data collection All data from the baseline and final evaluations were collected through the Zoom app or by WhatsApp video call and using survey monkey.

Primary response variable: physical performance

Physical performance was assessed with the short physical performance battery (SPPB) scale which is an instrument that evaluates three domains of physical performance: balance, gait speed, and lower limb strength to rise from a chair. Every test has a maximum score of 4, obtaining a maximum score of 12 points, if the subject obtains a score ≤ 8 points is classified as a person with low physical performance according to Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2).

Covariates

Sociodemographic: Age (years), sex, and schooling (<10; ≥10 years).Health Conditions: depressive symptoms were evaluated by the Depression Scale of the Center for Epidemiological Studies (CESD-7), cognitive status was assessed using the MMSE test , comorbidity through the Charlson comorbidity index , frailty was measured using the FRAIL scale (a simple frailty questionnaire), sarcopenia using the SARC-F scale (a screening questionnaire for sarcopenia) and medication use. It also evaluated functional disability (FD) using the Barthel scale for the basic activities of daily living (BADL) and the instrumental activities of daily living (IADL). Nutrition variables: malnutrition was assessed through the Mini Nutritional Assessment (MNA) test, anthropometric measurements such as weight (kg), height (mts), BMI (body mass index), calf, waist, hip and mild-arm circumferences, and body composition as fat mass (%) and free fat mass (%). These measurements were evaluated with an OMRON HBF-514C® portable scale capable of assessing a total weight of 150 kg. Level of physical activity: physical activity was measured using the Physical Activity Survey (YPAS) questionnaire, obtaining weekly METs as a result.

ELIGIBILITY:
The inclusion criteria were the following:

* Adults 60 and over years
* Adults who had an electronic device with internet access for video calls.

The exclusion criteria were:

* Adults self-reported walking disability, with the inability to complete the short physical performance battery (SPPB)
* Adults with severe functional dependence (defined as a Barthel index ≤ 60/100 score)
* Adults with cognitive impairment (defined as a mini-mental state examination (MMSE) score <24/30)
* Adults with terminal illness
* Adults who were participating in a physical activity or nutritional program
* Adults with a limb loss or use of lower or upper limb prostheses
* Adults with a history of injuries (fractures/falls) of less than one year in hip, knee or ankle joints and with surgery in the last 6 months or contraindications to perform trial activities in the judgment of medical personnel.
* Adults who presented any medical condition or adverse symptoms during the intervention that made it impossible to carry out the physical exercise program
* Adults who did not keep three times consecutive were eliminated from the study.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The participants were randomly selected regardless of gender
Enrollment: 110 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Physical performance | 3 months
  Physical performance was assessed with an short battery physical performance which is an instrument that evaluates three domains of physical performance: balance, gait speed, and lower limb strength to rise from a chair.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Teresa López Teros, PhD, Principal Investigator — Universidad Iberoamericana, A.C.
Locations (1):
- Iberoamerican University, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be used only for research purposes and the personal data of all participants will be respected.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The information will be protected by the principal investigator
Access Criteria: The information will only be shared with co-investigators of the project and for research purposes.